CLINICAL TRIAL: NCT04475536
Title: A Prospective Study, Single-arm, Multicentre, Observational to Evaluate Safety and Effectiveness of Stent Ultimaster Tansei Coronary Stent in Complex Coronary Lesions.
Acronym: TANSEI
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC08-TANSEI
Record Dates: First submitted 2020-07-16; First posted 2020-07-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease
Keywords: Complex Lesions
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: TANSEI stent

INTERVENTIONS:
Device: TANSEI stent — stenting with the TANSEI sirolimus-eluting stent

SUMMARY:
This prospective registry is intended to evaluate the safety and efficacy of the TANSEI stent.

DETAILED DESCRIPTION:
This prospective registry is intended to analyze clinical outcomes in patients treated with TANSEI stent in patients with complex coronary lesions .

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* With indication of percutaneous revascularization.
* Complex coronary lesion defined as:

  * Left main lesion AND/OR
  * Lesion located at a major bifurcation (side branch >2mm) AND/OR
  * Lesion located in a small vessel (<2.5 mm reference diameter by visual estimation) AND/OR
  * Lesion length > 35 mm
* Informed consent signed.

Exclusion Criteria:

* Cardiogenic shock at the time of the PCI(Percutaneous Coronary Intervention).
* Life expectancy of the patient under 1 year.
* Patients included in other studies or clinical trials.
* Clinical decision that excludes the use of drug-eluting stents.
* Confirmed allergy to aspirin and / or thienopyridines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with de novo native and complex coronary artery lesions, candidate to undergo revascularisation with a coronary device.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Safety.The composite of cardiac death, myocardial infarction (MI) and stent thrombosis (Academic Research Consortium definitive/probable). | 12 months
  The composite of cardiac death, myocardial infarction (MI) and stent thrombosis (Academic Research Consortium definitive/probable).
Efficacy.The incidence of clinically driven target lesion revascularization. | 12 months
  The incidence of clinically driven target lesion revascularization (TLR).

SECONDARY OUTCOMES:
All death. | 12 months
  All death.
Cardiac death. | 12 months
  Cardiac death.
Target Vessel revascularization. | 12 months
  Target Vessel revascularization.
Target lesion revascularization. | 12 months
  Target lesion revascularization.
Stent thrombosis (ARC definite/probable). | 12 months
  Stent thrombosis (ARC definite/probable).
Major bleeding event (BARC type 2-5). | 12 months
  Major bleeding event (BARC type 2-5).
Stroke. | 12 months
  Stroke.
Procedural success. | 12 months
  Procedural success ( Residual stenosis <30% after implantation at the narrowest point of the treated vascular segment).
Rate of patients with DAPT | From 1 to 6 months
  Rate of patients with DAPT
Rate of patients with DAPT | From 6 to 12 months
  Rate of patients with DAPT

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, LA Coruña
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General Universitario, Albacete
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital General Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Clinico Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Marques de Valdcilla, Santander
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Background] Saito S, Valdes-Chavarri M, Richardt G, Moreno R, Iniguez Romo A, Barbato E, Carrie D, Ando K, Merkely B, Kornowski R, Eltchaninoff H, James S, Wijns W; CENTURY II Investigators. A randomized, prospective, intercontinental evaluation of a bioresorbable polymer sirolimus-eluting coronary stent system: the CENTURY II (Clinical Evaluation of New Terumo Drug-Eluting Coronary Stent System in the Treatment of Patients with Coronary Artery Disease) trial. Eur Heart J. 2014 Aug 7;35(30):2021-31. doi: 10.1093/eurheartj/ehu210. Epub 2014 May 19. PMID 24847155
- [Background] Orvin K, Carrie D, Richardt G, Desmet W, Assali A, Werner G, Ikari Y, Fujii K, Goicolea J, Dangoisse V, Manari A, Saito S, Wijns W, Kornowski R. Comparison of sirolimus eluting stent with bioresorbable polymer to everolimus eluting stent with permanent polymer in bifurcation lesions: Results from CENTURY II trial. Catheter Cardiovasc Interv. 2016 May;87(6):1092-100. doi: 10.1002/ccd.26150. Epub 2015 Aug 13. PMID 26268482
- [Background] Lesiak M, Araszkiewicz A, Grajek S, Colombo A, Lalmand J, Carstensen S, Namiki A, Tobaru T, Merkely B, Moreno R, Barbato E, Wijns W, Saito S. Long Coronary Lesions Treated With Thin Strut Bioresorbable Polymer Drug Eluting Stent: Experience From Multicentre Randomized CENTURY II Study. J Interv Cardiol. 2016 Feb;29(1):47-56. doi: 10.1111/joic.12262. PMID 26864951
- [Background] Derimay F, Souteyrand G, Motreff P, Rioufol G, Finet G. Influence of platform design of six different drug-eluting stents in provisional coronary bifurcation stenting by rePOT sequence: a comparative bench analysis. EuroIntervention. 2017 Oct 13;13(9):e1092-e1095. doi: 10.4244/EIJ-D-16-00863. PMID 28485275
- [Background] Chevalier B, Smits PC, Carrie D, Mehilli J, Van Boven AJ, Regar E, Sawaya FJ, Chamie D, Kraaijeveld AO, Hovasse T, Vlachojannis GJ. Serial Assessment of Strut Coverage of Biodegradable Polymer Drug-Eluting Stent at 1, 2, and 3 Months After Stent Implantation by Optical Frequency Domain Imaging: The DISCOVERY 1TO3 Study (Evaluation With OFDI of Strut Coverage of Terumo New Drug Eluting Stent With Biodegradable Polymer at 1, 2, and 3 Months). Circ Cardiovasc Interv. 2017 Dec;10(12):e004801. doi: 10.1161/CIRCINTERVENTIONS.116.004801. PMID 29246909